CLINICAL TRIAL: NCT04524260
Title: Postoperative Outcome After the Application of Perioperative Painting Art Therapy (LOM® Solution Centered Art Therapy) in Patients Undergoing Major Surgery at the University Hospital of Zurich
Brief Title: The Effects of Perioperative Painting Art Therapy (LOM® Solution Centered Art Therapy) in Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAINT - Zurich; 2019-00643 (Other: Cantonal Ethics Committee Zurich); SNCTP000003688 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2020-03-19; First posted 2020-08-24 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Lower Gastrointestinal Neoplasms Benign; Pancreas Cancer; Posttraumatic Stress Disorder; Depression, Anxiety
Keywords: painting art therapy; PTSD; alternative/complementary medicine; anxiety
MeSH Terms: conditions — Pancreatic Neoplasms; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painting art therapy (Active Comparator): Intervention group
  Interventions: Behavioral: perioperative painting art therapy (LOM® solution centered art therapy)
- Usual Care (Sham Comparator): Control group
  Interventions: Behavioral: perioperative painting art therapy (LOM® solution centered art therapy) - control

INTERVENTIONS:
Behavioral: perioperative painting art therapy (LOM® solution centered art therapy) — We plan to apply painting art therapy as a health-related intervention to patients coming to our department for elective major surgery of the pancreatic and lower gastrointestinal tract for malignant pathologies. Patients will have 3 patient art therapy sessions: one before surgery, one on day 3-5 after surgery during the hospital stay and one during the follow-up 6 weeks postoperative
  Arms: Painting art therapy
Behavioral: perioperative painting art therapy (LOM® solution centered art therapy) - control — "usual care", no particular intervention during the perioperative setting. There will be 2-3 painting art therapy sessions after the follow-up 6 weeks postoperative. Therefore this group is called "usual care"- or delayed intervention group.
  Arms: Usual Care

SUMMARY:
The investigators want to study whether the use of painting art therapy has an influence on the quality of life, the complication rate and the general outcome of major abdominal surgery. The painting art therapy is carried out according to the protocol of (LOM® Solution Centered Art Therapy) by trained painting art therapists.

DETAILED DESCRIPTION:
The interest in alternative and complementary medical treatments has increased significantly in recent years and several studies showed a positive effect on the healing process of patients undergoing surgery. Painting art therapy represents another possible form of such a complementary medical treatment. However, the effect in the context of major abdominal surgical interventions has not yet been investigated, which is why the investigators are conducting this study. Selected patients referred to the Department of Visceral and Transplantation Surgery with operable pathologies of the pancreatic and the lower gastrointestinal tract are subjected to perioperative painting art therapy. It is carried out according to the protocol of (LOM® Solution Centered Art Therapy) by trained painting art therapists. The investigators want to evaluate the effectiveness of perioperative painting art therapy by analyzing the results of several questionnaires regarding anxiety and depression levels as well as health related patient data to observe the short/long term outcome and the psychological well-being of patients undergoing major surgery in case of carcinoma. The aim of the study is to assess if painting art therapy, more precisely the LOM®-method, is effective in reducing symptoms of anxiety and depression in patients undergoing surgery. When it appears that the application of perioperative painting art therapy has a major influence on the postoperative outcome in cancer patients, some patients could benefit from a noninvasive, low-risk and easy additional treatment option. This study is a collaboration with the Institute of Complementary and Integrative medicine of the University Hospital Zurich.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients of both genders ≥ 18 years subjected to major (oncological) surgery due to pathologies of the pancreatic and lower gastrointestinal tract at our department.
* The initial diagnosis does not date back longer than 6 months prior the planned surgery. Neoadjuvant radio-/chemotherapy is not an exclusion criteria.
* Able to speak and understand German or English
* Signed written informed consent by the participant after extensive oral and written information about the research project and its aims.
* Thresholds of primary outcome: anxiety levels measured with STAI-form Y-1 (state) and Y-2 (trait). Thresholds: scores between 20 (minimum) and 80 (maximum) in each subscore.

Exclusion Criteria:

* Woman who are pregnant or breast feeding.
* Known or suspected non-compliance regarding the execution of painting art therapy and/or the proper completion of the needed forms.
* Drug or alcohol abuse.
* Regular intake of antidepressant medication with the exception of medication prescribed for chronic insomnia.
* Acute suicidality.
* Life expectancy less than 9 months after planned surgery.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, ect. of the participant
* Participation in another study during the present study and within 6 weeks following the surgery.
* Previous enrollment into the current study.
* Enrollment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of Anxiety | Change from Baseline STAI-Score up to 6 months post surgery
  State Trait Anxiety Inventory, STAI-forms Y-1/state and Y-2/trait (questionnaire), scores range from 20 to 80, with higher scores correlating with greater anxiety

SECONDARY OUTCOMES:
Change of Depression | Change from Baseline PHQ-9-Score up to 6 months post surgery
  PHQ-9 ("Brief Patient Health Questionnaire-9"), scores ranging from 0 to 27, with higher scores correlating with greater depression
Change of Quality of Life - PROMIS 29 | Change from Baseline PROMIS 29-Scores up to 6 months post surgery
  PROMIS 29 ("Profile Physical and Mental Health Summary Scores"-questionnaire), scores ranging from 28 to 150, with higher scores correlating with lower quality of life
Change of Health related quality of life - SF-12 | Change from Baseline SF-12-Scores up to 6 months post surgery
  SF-12 ("short form 12", 12 question survey), results calculated with scoring programme, with higher scores correlating with lower quality of life

OTHER OUTCOMES:
Change of Postoperative Pain 1 | Change from Baseline (NRS pain 0-10) at 6 months post surgery
  Subjectively perceived (NRS 0-10)
Change of Postoperative Pain 2 | Change from Baseline (amount of analgesia) at 6 months post surgery
  Amount of Analgesia (data)
Change of Blood pressure | Change from Baseline at 6 months post surgery
  Systolic and diastolic BP in mmHg
Change of Heart Rate | Change from Baseline at 6 months post surgery
  HR in bpm (beats per minute)
Change of Respiratory Rate | Change from Baseline at 6 months post surgery
  RR/min
Laboratory result, chemistry (CRP) | Change from Baseline at 6 months post surgery
  C-reactive protein (mg/l)
Laboratory result, hematology (Hb) | Change from Baseline at 6 months post surgery
  Hemoglobin, measured in g/l
Laboratory result, hematology (Leucocytes, White Blood Cells) | Change from Baseline at 6 months post surgery
  WBCs measured in G/l
Complications (Clavien-Dindo-Classification) | 6 months
  Clavien-Dindo-Classification (classified from 0 - V), higher numbers according to more severe complications, V is dead)
Complications (CCI during hospital stay) | 6 months
  CCI during hospital stay; measured from healthy (0) to death (100)
Tumor staging assessed according official TNM-Staging | 1 week postoperative (as soon as final histopathology is available)
  TNM-Classification of Malignant Tumors, 8th edition
Socio-economic: days in hospital | up to 6 months post surgery
  Days in hospital until discharge, measured in days
Socio-economic: days in ICU | up to 6 months post surgery
  Days in ICU until discharge to regular unit, measured in days
Socio-economic: ability to return to work | up to 6 months post surgery
  Measured will be the time from surgery until return to work, in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alain Clavien, MD PhD, Study Chair — Department of Visceral- and Transplantation Surgery, University Hospital Zurich
Locations (1):
- Department of Visceral- and Transplantation Surgery, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No